CLINICAL TRIAL: NCT03936348
Title: Evaluation of a Respiratory Muscle Training Program Restricting Nasal Breathing With FeelBreathe® Device in COPD Patients
Brief Title: Effects of an Exercise Rehabilitation Programme With a Nasal Inspiratory Restriction Device in COPD Patients
Acronym: EPOC_2_0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other); Hospital Universitario Puerta del Mar (Other); Bahía Sur Andalusian Center for Sports Medicine (Unknown)
Responsible Party: Principal Investigator, Jesus Gustavo Ponce González, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: (SEPAR): CÓDIGO: 099/2015
Record Dates: First submitted 2019-04-28; First posted 2019-05-03 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Breathing Exercises; Exercise Tolerance
Keywords: Pulmonary rehabilitation; Medical device; FeelBreathe; Exercise intervention; Equipment and Supplies
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients were randomized to 3 groups. The first one performed a supervised RP using the Feelbreathe® device (FB group), the second group developed the same RP with oronasal breathing without FB (ONB group) and the third was the control group (CG). The RP was conducted during 8 weeks, 3 days per week, and includes a combined training of endurance and strength exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FB group (Experimental): Participants who performed an exercise training program for 8 weeks using a nasal restriction device for inspiratory muscle training, called Feelbreathe®
  Interventions: Device: Exercise training program with and without FB
- ONB group (Experimental): Participants who performed an exercise training program for 8 weeks with oronasal breathing without FB
  Interventions: Device: Exercise training program with and without FB
- control group (CG) (No Intervention): Participants who received the standard medical recommendations for patients with COPD, but not participated in the exercise intervention program

INTERVENTIONS:
Device: Exercise training program with and without FB — Participants carried out a supervised RP for 8 weeks, 3 days per week. The training sessions lasted 60 minutes and included a warning up phase, the main phase and a recovery phase. After each session, Borg's perceived exertion was measured. The Rehabilitation Program (RP) included aerobic exercise on cycle ergometer and on treadmill (progressing since 10' to 30' and since 40 to 75% of the reserve heart rate (RHR) or 6-7 score based on Borg's perceived exertion), strengthening of lower and upper limb muscles groups, breathing exercises (pursed lip breathing, diaphragmatic and abdominal breathing and diaphragmatic mobility) and finally stretching exercises.
  In the FB group, for restricted nasal breathing, at the beginning of the training program, the small size device was used (4 mm). The size of the device was progressively increasing according to the patient adaptation to the 5 or 6 mm device, depending on the score on Borg's perceived exertion scale.
  Other Names: Pulmonary rehabilitation program
  Arms: FB group; ONB group

SUMMARY:
This study evaluates the effects of a nasal restriction device for inspiratory muscle training (FeelBreathe) after 8 weeks of exercise intervention on exercise capacity, quality of life, dyspnea and inspitarotory muscle strength in patients with stable COPD. Participants were divided in three groups: 1) exercise intervention using the Feelbreathe® device (FB group), 2) exercise intervention with oronasal breathing without FB (ONB group) and 3) no participation in the exercise intervention as control group (CG).

DETAILED DESCRIPTION:
The Feelbreathe® device, tested in the investigator's study can be used in static and dynamic situations and is a nasal ventilatory flow restriction device made by a strip of hypoallergenic material (3M Spain, S.A. Medical Specialties / O.E.M.) that is placed and adhered under the nostrils impairing the free pass of air through the nose by producing resistance to flow. Depend on the size or/and porosity of the device, the inspiratory process is more or less difficult. It can be used while performing dynamic exercise or doing daily living activities. The Feelbreathe® device (FB) has been authorized by the Spanish Agency for Medicines and Health Products for application on COPD patients (Expedient 521/15/EC. AEMPS-Madrid-Spain-Patent Nº: P200902402).

ELIGIBILITY:
Inclusion Criteria:

* men with diagnosis of COPD according to guidelines criteria
* with moderate or severe airflow obstruction (GOLD 2 or 3)
* dyspnea grade 2 or greater by mMRC scale
* stable clinical condition for at least 2 months.

Exclusion Criteria:

* poor compliance
* treatment with oxygen therapy or non-invasive mechanical ventilation
* CO2 retention
* medical conditions that can produce or increase dyspnea on exercise in addition to COPD (cardiovascular, metabolic or other respiratory diseases)
* osteoarticular or neuromuscular diseases that may limit the correct performance of the 6MWT

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake during incremental test to exhaustion on treadmill | 8 WEEKS
  mL/min
Ventilation during incremental test to exhaustion on treadmill | 8 WEEKS
  L/min

SECONDARY OUTCOMES:
dyspnea scale | 8 WEEKS
  mMRC (Modified Medical Research Council) Dyspnea Scale. Values from 0 (better) to 4 (worse) about disability attributable to breathlessness
The COPD Assessment Test (CAT) is a questionnaire for people with Chronic Obstructive Pulmonary Disease (COPD) | 8 WEEKS
  The COPD Assessment Test (CAT) score measures the impact that COPD (Chronic Obstructive Pulmonary Disease) is having on the wellbeing and daily life of the patient. Score from 0 (better) to 40 (worse) about the impact of COPD symptoms on patients' overall health.
exercise capacity using the distance walked in the six minutes walking test (6MWT) | 8 WEEKS
  distance measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Jose L González Montesinos, PhD, Principal Investigator — University of Cádiz

IPD SHARING:
Plan to Share IPD: No
Since there is personal and not transferable data

REFERENCES:
- [Background] González-Montesinos JL, Vaz Pardal C, Fernández Santos JR, Arnedillo Muñoz A CSJ y GE de los MR. Efectos del entrenamiento de la musculatura respiratoria sobre el rendimiento. Revisión bibliográfica. Rev Andal Med Deport. 2012;5(4):163-70.
- [Result] González Montesinos JL, Costa Sepúlveda JL, Fernández Santos J, Gómez Espinosa de los Monteros R, Mora Vicente J, Castro Piñero J y, et al. Dispositivo de Restricción y Filtrado del Flujo Ventilatorio Nasal. P200902402, 2011. p. 1-4.
- [Result] Gonzalez-Montesinos JL, Ponce-Gonzalez JG, Vicente-Campos D, Lopez-Chicharro J, Fernandez-Santos Jdel R, Vaz-Pardal C, Costa-Sepulveda JL, Conde-Caveda J, Castro-Pinero J. Efectos de un dispositivo de restriccion ventilatoria nasal sobre la ventilacion pulmonar e intercambio gaseoso durante el ejercicio en personas sanas. Nutr Hosp. 2016 Mar 25;33(2):130. doi: 10.20960/nh.130. PMID 27238811
- [Result] Scherer TA, Spengler CM, Owassapian D, Imhof E, Boutellier U. Respiratory muscle endurance training in chronic obstructive pulmonary disease: impact on exercise capacity, dyspnea, and quality of life. Am J Respir Crit Care Med. 2000 Nov;162(5):1709-14. doi: 10.1164/ajrccm.162.5.9912026. PMID 11069801
- [Result] Wada JT, Borges-Santos E, Porras DC, Paisani DM, Cukier A, Lunardi AC, Carvalho CR. Effects of aerobic training combined with respiratory muscle stretching on the functional exercise capacity and thoracoabdominal kinematics in patients with COPD: a randomized and controlled trial. Int J Chron Obstruct Pulmon Dis. 2016 Oct 28;11:2691-2700. doi: 10.2147/COPD.S114548. eCollection 2016. PMID 27822031
- [Result] Camillo CA, Osadnik CR, van Remoortel H, Burtin C, Janssens W, Troosters T. Effect of "add-on" interventions on exercise training in individuals with COPD: a systematic review. ERJ Open Res. 2016 Mar 29;2(1):00078-2015. doi: 10.1183/23120541.00078-2015. eCollection 2016 Jan. PMID 27730178

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03936348/Prot_SAP_000.pdf